CLINICAL TRIAL: NCT04194320
Title: Nalbuphine Versus Dexamethasone as an Adjuvant to Lidocaine / Bupivacaine Mixture in Ultrasound-guided Supraclavicular Brachial Plexus Block for Upper Limb Surgeries
Brief Title: Dexamethasone Versus Nalbuphine as Adjuvants in Brachial Plexus Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Brachial Plexus Block
Record Dates: First submitted 2019-12-08; First posted 2019-12-11 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2020-07

CONDITIONS: Anesthesia
MeSH Terms: interventions — High-Energy Shock Waves

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group I "Placebo" (Placebo Comparator): Ultrasound (US) guided supraclavicular brachial plexus block will be done to the patients who are prepared to undergo upper limb surgeries below the level of the shoulder within the distribution of supraclavicular brachial plexus block using: 30 mL volume of local anesthetics (Lidocaine 2% + bupivacaine 0.5% 1:1 mixture) + 2 ml 0.9% normal saline.
  Interventions: Procedure: Ultrasound (US) guided supraclavicular brachial plexus block
- Group II "Nalbuphine " (Active Comparator): Ultrasound (US) guided supraclavicular brachial plexus block will be done to the patients who are prepared to undergo upper limb surgeries below the level of the shoulder within the distribution of supraclavicular brachial plexus block using: 30 mL volume of local anesthetics (Lidocaine 2% + bupivacaine 0.5% 1:1 mixture) + 10 mg nalbuphine hydrochloride (completed to 2 ml with 0.9% normal saline).
  Interventions: Procedure: Ultrasound (US) guided supraclavicular brachial plexus block
- Group III "Dexamethasone" (Active Comparator): Ultrasound (US) guided supraclavicular brachial plexus block will be done to the patients who are prepared to undergo upper limb surgeries below the level of the shoulder within the distribution of supraclavicular brachial plexus block using: 30 mL volume of local anesthetics (Lidocaine 2% + bupivacaine 0.5% 1:1 mixture) + 2 mL dexamethasone 0.4% (8 mg).
  Interventions: Procedure: Ultrasound (US) guided supraclavicular brachial plexus block

INTERVENTIONS:
Procedure: Ultrasound (US) guided supraclavicular brachial plexus block — Using 8 mg dexamethasone or 10 mg nalbuphine as adjuvants to (Lidocaine 2% + bupivacaine 0.5% 1:1 mixture) in ultrasound (US) guided supraclavicular brachial plexus block

SUMMARY:
Brachial plexus block is a very reliable method of regional anesthesia for the upper limb. It achieves ideal operating conditions by producing complete muscular relaxation and stable intraoperative hemodynamics.However,Local anesthetics alone have a shorter duration of postoperative analgesia. Hence,various adjuvants have been added to local anesthetics to achieve quick, dense, and prolonged block. This study assess and compare the efficacy of dexamethasone or nalbuphine as adjuvants to local anesthetics in supraclavicular brachial plexus block for upper limb surgeries.

DETAILED DESCRIPTION:
Upper-limb surgeries can be performed under either general or regional anesthesia.However, regional anesthesia has the advantages of long-lasting pain relief & avoidance of airway instrumentation.Brachial plexus block is a very reliable method of regional anesthesia for the upper limb. It achieves ideal operating conditions by producing complete muscular relaxation and stable intraoperative hemodynamics.However,Local anesthetics alone have a shorter duration of postoperative analgesia. Hence,various adjuvants have been added to local anesthetics to achieve quick, dense, and prolonged block. This study assess and compare the efficacy of using 8 mg dexamethasone or 10 mg nalbuphine as adjuvants to local anesthetics mixture (Lidocaine 2% + bupivacaine 0.5% 1:1 mixture) in Ultrasound-guided supraclavicular brachial plexus block for upper limb surgeries below the level of the shoulder.

ELIGIBILITY:
Inclusion Criteria:

* Patient acceptance.
* American Society of Anesthesiologists (ASA) I and (ASA) II.
* Age 21-60 years old.
* Both gender.
* BMI < 30.
* Accepted mental state of the patient.
* Unilateral upper limb surgeries below the level of the shoulder.

Exclusion Criteria:

* Patient refusal.
* Peripheral neuropathy.
* Pathological coagulopathy.
* Infection at the injection site.
* History of active substance abuse.
* Untreated pneumothorax.
* Disturbed conscious level.
* An allergy to local anesthetics or nalbuphine or dexamethasone.
* Planned for receiving general anesthesia during the same operation for any cause.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2020-05-05 (Actual); Study Completion 2020-06-15 (Actual)

PRIMARY OUTCOMES:
Duration of postoperative analgesia | First 24 hours after surgery
  Time between onset of sensory block to the first report of postoperative pain at the surgical site that has a VAS "visual analogue score" ≥ 4.

SECONDARY OUTCOMES:
post operative pain score "Visual Analogue Score" | First 24 hours after surgery
  On a scale of 0-10, the patient will be asked to quantify postoperative pain as the following: 0: No pain 10: Maximum/worst imaginable pain. Visual Analog Scale assessment will be done every 5 minutes for first 30 minutes, then hourly for first 8 hours then every 4 hourly till patient complained of pain equivalent to a VAS score of 4. Rescue analgesia (injection of fentanyl 25 mcg intravenous increments) up to 200 μg/hour is administered when VAS score reached 4.
The total opioid consumption | First 24 hours after surgery
  Total dose of fentanyl as a rescue analgesic in the first 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed ELSayed, MSc, Principal Investigator — Faculty of medicine, zagazig university, Egypt; Ahmed mohamed Salama, MD, Study Chair — Faculty of medicine, zagazig university, Egypt; Ayman Abd-El Salam Hassan, MD, Study Chair — Faculty of medicine, zagazig university, Egypt; Fatma Mahmoud Ahmed, MD, Study Director — Faculty of medicine, zagazig university, Egypt
Locations (1):
- Faculty of medicine, Zagazig University, Zagazig, Al-Sharkia, Egypt

REFERENCES:
- [Background] Abdallah FW, Johnson J, Chan V, Murgatroyd H, Ghafari M, Ami N, Jin R, Brull R. Intravenous dexamethasone and perineural dexamethasone similarly prolong the duration of analgesia after supraclavicular brachial plexus block: a randomized, triple-arm, double-blind, placebo-controlled trial. Reg Anesth Pain Med. 2015 Mar-Apr;40(2):125-32. doi: 10.1097/AAP.0000000000000210. PMID 25629321
- [Background] Das A, RoyBasunia S, Mukherjee A, Biswas H, Biswas R, Mitra T, Chattopadhyay S, Mandal SK. Perineural Nalbuphine in Ambulatory Upper Limb Surgery: A Comparison of Effects of Levobupivacaine with and without Nalbuphine as Adjuvant in Supraclavicular Brachial Plexus Block - A Prospective, Double-blinded, Randomized Controlled Study. Anesth Essays Res. 2017 Jan-Mar;11(1):40-46. doi: 10.4103/0259-1162.200225. PMID 28298754
- [Background] Perlas A, Lobo G, Lo N, Brull R, Chan VW, Karkhanis R. Ultrasound-guided supraclavicular block: outcome of 510 consecutive cases. Reg Anesth Pain Med. 2009 Mar-Apr;34(2):171-6. doi: 10.1097/AAP.0b013e31819a3f81. PMID 19282715